CLINICAL TRIAL: NCT00382902
Title: Clinical Evaluation of the Safety and Efficacy of an Investigational Multi-Purpose Disinfecting Solution Compared to Two Marketed Multi-Purpose Solutions for Care of Silicone Hydrogel Soft Contact Lenses
Brief Title: Evaluation of an Investigational Multi-Purpose Disinfecting Solution for the Care of Silicone Hydrogel Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-13
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2006-09

CONDITIONS: Contact Lens Care
Keywords: Contact Lens Care

INTERVENTIONS:
Device: OptiFree Multi-Purpose Disinfecting Solution

SUMMARY:
The objective of the study was to clinically evaluate the safety and effectiveness of a new multi-purpose disinfecting solution in patients wearing silicone hydrogel soft contact lenses.

ELIGIBILITY:
* Successful daily wear of Night & Day® or Acuvue® Advance™ silicone hydrogel contact for at least two weeks.
* Use of AOSEPT® ClearCare™ only as the pre-study care regimen for at least two weeks (rewetting drops use is also acceptable).
* Successful lens wear for at least 8 hours per day.
* Vision correctable to 20/30.
* Normal eyes - no current ocular abnormalities that prevent successful contact lens wear.
* No corneal surgery within the past 12 months.
* No systemic disease that affects that eye or that could be worsened by the use of contact lenses or solutions.
* No over-the-counter or prescription ocular medication.
* No enrollment in another clinical study within 30 days prior to enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 233
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining (Type and Area)
Conjunctival Staining
Lens Deposits
Subject Questions/Subject Likert Questionnaire
Ocular Comfort and Symptom Scales
Lens Replacement Incidence and Causality
Corrected Visual Acuity with Study Lenses (Snellen)
Average Lens Wearing Time
Average Uncomfortable Lens Wearing Time
Safety:
Slit-lamp Findings - Cornea: Edema, Neovascularization, Infiltrates; Injection, Tarsal Abnormalities and Other Complications
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Napier, Study Director — Alcon Research
Locations (1):
- Portland Site, Portland, Maine, United States